CLINICAL TRIAL: NCT05116683
Title: A Phase II Study, With a Safety lead-in, to Evaluate ATX-101, a Peptide Drug Targeting PCNA, in Advanced Dedifferentiated Liposarcoma and Leiomyosarcoma
Brief Title: ATX-101 in Advanced Dedifferentiated Liposarcoma and Leiomyosarcoma
Acronym: ATX-101
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by PI
Sponsor: Benjamin Izar (Other)
Responsible Party: Sponsor-Investigator, Benjamin Izar, Assistant Professor, Division of Hematology/Oncology, Department of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT7079
Record Dates: First submitted 2021-10-18; First posted 2021-11-11 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Leiomyosarcoma; Liposarcoma
Keywords: LMS; LPS; ATX-101
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATX-101 (Experimental): Patients will be treated with ATX-101 60 mg/m2 IV weekly in continuous 21 day cycles. Patients will receive premedication prior to the ATX-101 infusion to reduce the risk of infusion-related reactions.
  Interventions: Drug: ATX-101

INTERVENTIONS:
Drug: ATX-101 — Patients will be given ATX-101 at 60 mg/m2 IV weekly in continuous 21 day cycles.
  Other Names: ATX-101 drug substance

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a new investigational drug, ATX-101, for the treatment of dedifferentiated liposarcoma (LPS) and leiomyosarcoma (LMS). ATX-101 is an intravenous (IV) drug which blocks the interaction of a protein called PCNA with a number of "stress response" proteins. These interactions are thought to be important for cancer cell survival and growth. ATX-101 may disrupt these interactions and therefore help treat the cancer. In this study, all patients will receive the same treatment. Most of the exams, tests, and procedures are part of the usual approach to medical care for this condition. However, some additional tests or procedures may be performed, and other tests may be performed more frequently than usual.

DETAILED DESCRIPTION:
ATX-101 is a small molecule peptide comprised of a novel human proliferating cell nuclear antigen (PCNA) interacting motif termed APIM coupled to cellular and nuclear delivery domains. PCNA interacts with many cellular proteins and exerts pleiotropic effects in the cancer cell. Proteins that bind to PCNA via APIM are especially important in the cellular stress and DNA damage responses, as well as intracellular signaling, apoptosis, metabolism and anti-tumor immunity. In preclinical studies, ATX-101 demonstrated single-agent activity and potentiated other cytotoxic and targeted agents across multiple cancer models in vitro and in vivo, including LMS and LPS. ATX-101 is currently being evaluated in a phase 1 safety and pharmacokinetic study in solid tumors using a 3 + 3 dose escalation design. As of 10/29/2020, ATX-101 has been evaluated across dose levels of 20 mg/m2 - 60 mg/m2 IV weekly. Although no maximum tolerated dose (MTD) was reached, after review of the available safety data, the RP2D was determined to be 60 mg/m2 IV weekly, with no plans to dose escalate further. ATX-101 has been well tolerated, with no grade 3 or higher adverse events (AEs) observed during the phase 1 study. Common AEs include grade 1/2 infusion related reactions (which have been easily managed with supportive care), mild fatigue and diarrhea. In this study, ATX-101 demonstrated encouraging activity as prolonged disease stabilization in patients with progressive, heavily pre-treated malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed dedifferentiated liposarcoma (LPS) or leiomyosarcoma
* ATX-101 in Sarcoma Phase II
* (LMS). Pathology review occurs at the center enrolling the patient on this trial.
* Disease must be locally advanced and unresectable or metastatic. Disease which may be resected but with an associated level of morbidity deemed unacceptable by the treating clinician is considered eligible.
* Patients must have measurable disease by RECIST criteria version 1.1. In addition, the first 10 patients enrolled on the study must have a site of disease amenable to image-guided biopsy at minimal risk or less, and must agree to undergo this biopsy.
* Patients must evidence of disease progression, either clinically or radiographically, within the 12 weeks prior to study enrollment, as determined by the investigator enrolling the patient on the study.
* Patients must have been treated with at least one prior systemic regimen for advanced sarcoma: LMS: Anthracycline-based chemotherapy, or gemcitabine/docetaxel. LPS: No specification as to the prior treatment received. Neoadjuvant or adjuvant systemic therapy does not qualify as prior treatment unless completed within 6 months of disease relapse.
* Patients must be age 18 years or older. Because the safety of ATX-101 in patients less than 18 years of age has not been characterized, children are excluded from the present study.
* Patients must demonstrate an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Patients must demonstrate normal organ and marrow function as defined below:
* Absolute neutrophil count (ANC) ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Creatinine ≤ 1.5 times upper limit of normal OR
* Calculated creatinine clearance > 45 mL/min*
* Total bilirubin ≤ 1.5 times upper limit of normal**
* Aspartate transaminase (AST)/aminotransferase (ALT) ≤ 1.5 times upper limit of normal**
* Notes: Upper limit of normal is defined by the clinical laboratory performing the test.
* Using the lean body mass formula only (Modified Cockcroft Gault) ** If transaminase elevation and/or bilirubin elevation is attributed to the presence of liver metastases, a total bilirubin ≤ 2.5 times the upper limit of normal and an AST and ALT ≤ 2.5 times the upper limit of normal are permissible. Patients with an elevated bilirubin level that is attributed to an inherited disorder, such as Gilbert's disease, may be enrolled at the discretion of the principal investigator.
* The effects of ATX-101 on the developing human fetus are unknown. For this reason, women of child-bearing potential and all men must agree to use adequate contraception (for women: hormonal or barrier method of birth control, abstinence; for men: male condom, prior vasectomy, or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ATX-101 administration. If patients do not agree to the above, they are not considered eligible.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria

* Patients must not have received treatment with any chemotherapy, immunotherapy, radiotherapy or an investigational agent for malignancy within the 21 days of initiating treatment on this protocol.
* Patients may not have received treatment with a small molecule targeted agent (including off-label or investigational use) within 14 days of initiating treatment on this protocol, provided this represents at least 7 half-lives for that agent.
* Toxic effects from any prior therapy (except alopecia) must have resolved to grade 1 or less according to NCI CTCAE v4.0 or to the patient's baseline by the time of initiating treatment on this protocol.
* Patients may not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, cerebrovascular accident within the last six months, uncontrolled diabetes mellitus, uncontrolled psychiatric illness or any other disease condition that would limit compliance with study requirements in the opinion of the principal investigator.
* Patients may not be pregnant or nursing. Pregnant women are excluded from this study because the teratogenic effects of ATX-101 have not been adequately studied. A negative pregnancy test must be documented 7 days or less prior to initiating treatment on this protocol. Because there is an unknown but potential risk for adverse events to nursing infants secondary to treatment of the mother with ATX-101, breastfeeding must be discontinued prior to enrollment.
* Patients may not have known active hepatitis B or C infection. In patients with a history of hepatitis B or C infection, resolution of infection must be demonstrated by negative serology for hepatitis B surface antigen (HBsAg) and/or negative hepatitis C virus (HCV) RNA.
* Patients may not have uncontrolled HIV/AIDS infection. However, HIV positive patients on highly active retroviral therapy (HAART) with an undetectable viral load and CD4 T-cell count above 200 may participate.
* Anticipated requirement for surgery during the study period or major surgery within 3 weeks of initiating treatment.
* Active central nervous system (CNS) metastases or leptomeningeal involvement. Patients with known CNS metastases must have received definitive radiotherapy or surgery at least 4 weeks prior to initiating treatment with imaging demonstrating no progression of disease over this interval.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Izar, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATX-101
Started | 4
Completed | 0
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | ATX-101
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  18-49 years | 0
  50-59 years | 2
  60-69 years | 0
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Rate (PFR)
Description: The study will evaluate the preliminary efficacy of ATX-101 in advanced L-sarcomas (LMS, LPS) by measuring the PFR (progression free rate) at 12 weeks (PFR12). Progression evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (the appearance of one or more new lesions is also considered progression).
Time Frame: 12 weeks
Population: Three of four participants analyzed due to n=1 participant who expired prior to week 12 (stable disease at time of death).
Measure: Count of Participants; unit: Participants
Arm/Group | ATX-101
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Number of Adverse Events
Description: Counted per adverse event basis by grade as evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The higher the grade, the more severe the event.
Time Frame: Up to approximately 7 months
Measure: Number; unit: Adverse Events
Arm/Group | ATX-101
Number analyzed (Participants) | 4
Adverse Events
  Grade 1 | 13
  Grade 2 | 16
  Grade 3 | 4
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of patients whose cancer shrinks or disappears after treatment. This will be measured by the percentage of patients having a complete or partial response per RECIST Version 1.1. ORR = Complete Response (CR) + Partial Response (PR); CR defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm and PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to approximately 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | ATX-101
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Duration of the Response
Description: Duration of response is measured from the time the measurement criteria for an objective response is recorded until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Up to approximately 7 months
Population: Zero analyzed as zero participants demonstrated objective response.
Arm/Group | ATX-101
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Median time from start treatment until the time of progression or death.
Time Frame: Up to approximately 5 months
Measure: Median (Full Range); unit: months
Arm/Group | ATX-101
Number analyzed (Participants) | 4
months | 2.46 [1.28 to 5.19]

6. Secondary Outcome: Median Overall Survival (OS)
Description: Median time from start of treatment until the time of death from any cause.
Time Frame: Up to approximately 7 months
Measure: Median (Full Range); unit: Months
Arm/Group | ATX-101
Number analyzed (Participants) | 4
Months | 4.40 [2.53 to 6.64]

ADVERSE EVENTS:
Time Frame: Up to approximately 7 months
Description: Adverse event assessment conducted at each follow up visit (day 1, 8, and 15 of each cycle).
Arm/Group | ATX-101
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATX-101 (N=4)
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATX-101 (N=4)
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Blood bilirubin increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Generalized edema (General disorders) | 1
Infusion related reaction (General disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05116683/Prot_SAP_000.pdf